CLINICAL TRIAL: NCT03358303
Title: Effect of a Mobile Phone-based Telemonitoring Program on the Outcome of Heart Failure Patients After an Incidence of Acute Decompensation
Brief Title: Effects of Telemonitoring on the Outcome of Heart Failure Patients After an Incidence of Acute Decompensation
Acronym: Medly-AID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); MOUNT SINAI HOSPITAL (Other); North York General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-5887
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure
Keywords: telemonitoring; smartphone application
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Medly) (Experimental): Medly is a smartphone application allows heart failure (HF) patients to measure and record their daily weight, blood pressure (BP), heart rate, and self-reported symptoms. This monitoring information is then transmitted wirelessly to a data server where an algorithm is used to generate an alert to a healthcare provider as necessary. The patient also receives an automated self-care message based on their measurements and reported symptoms.
  Interventions: Device: Medly
- Control (No Intervention): Standard of care: Control groups will receive standard medical care when discharged from hospital, including discharge instructions, home medications as well as follow-up in a heart failure clinic or with a primary care doctor.

INTERVENTIONS:
Device: Medly — Medly will enable patients with HF to take clinically relevant physiological measurements with wireless home medical devices and to answer symptom questions on the smartphone. The measurements will be automatically and wirelessly transmitted to the mobile phone and then to a data server. Automated self-care instructions/messages will be sent to the patient based on the readings and reported symptoms. If there are signs of their status deteriorating, an alert will be sent to a clinician that is responsible for the particular chronic condition of concern. The clinicians will have all the relevant patient data sent to them and will be able to access (through a secure web portal) to view historical and trending data for their patients.
  Arms: Telemonitoring (Medly)

SUMMARY:
Heart failure is the most rapidly rising cardiovascular disease and has come to be recognized as a growing epidemic. Digital health interventions are the most recent iteration of an effort to promote individualized outpatient care through positive behaviour change theory. The UHN team has developed a highly automated and user-centered smartphone-based system, Medly, which allows for the telemonitoring of patients diagnosed with heart failure. The purpose of this study will be two-fold: 1) to determine if the introduction of Medly within two weeks of discharge will improve self-care management, quality of life, and clinical status, 2) to assess whether Medly will lead to a potential reduction in 30 day readmission rates amongst HF patients in the Toronto Central Local Health Integration Network (TC LHIN), without increasing the average length of stay or visits to the emergency department. These parameters will be measured as secondary outcomes.

DETAILED DESCRIPTION:
Heart failure is the most rapidly rising cardiovascular disease and has come to be recognized as a growing epidemic. Digital health interventions are the most recent iteration of an effort to promote individualized outpatient care through positive behaviour change theory. The UHN team has developed a highly automated and user-centered smartphone-based system, Medly, which allows for the telemonitoring of patients diagnosed with heart failure

Patients with heart failure will be provided with a smartphone and commercial home medical devices, such as a blood pressure monitor and weight scale. The measurements from the medical devices will be automatically sent to the smartphone, and from there to a data server at the hospital for analysis and storage. Both clinicians and patients will be able to access these data and will be sent alerts by the system if the measurements are outside of the normal range. The system will be evaluated through interviews and comparing outcomes between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Hospitalization for decompensated HF > 48 hours
* Patient speaks and reads English adequately to provide informed consent and understand the text prompts in the application (or has an informal caregiver who can translate for them)
* Ability to comply with using Medly (ex. able to stand on the weight scale, able to answer symptom questions, etc.)

Exclusion Criteria:

* Dementia or uncontrolled psychiatric illness
* Residents of long-term care facilities
* Terminal diagnosis of any health condition with a life expectancy < 1 year
* Patients who will require inpatient rehabilitation after discharge
* Participating in another clinical trial that may confound the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-care of health failure | Baseline, 3 months
  Change in self-care of health failure as measured by the Self-Care of Heart Failure Index (SCHFI)
Change in quality of life | Baseline, 3 months
  Change in quality of life, as measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) and EuroQol (EQ5D)
Change BNP/NT-pro BNP levels | Baseline, 1 month, 3 months
  Change BNP/NT-pro BNP levels
Change in NYHA class | Baseline, 1 month, 3 months
  Change in NYHA class
Compliance with Medly utilization | 3 months
  Ability to adhere to Medly program

SECONDARY OUTCOMES:
Hospital length of stay | 0 - 3 months
  Hospital length of stay
30-day HF readmission rate | 1 month, 3 months
  30-day HF readmission rate
Number of visits to the emergency department | 0 - 3 months
  Number of visits to the emergency department

OTHER OUTCOMES:
Safety Endpoint: Change in creatinine levels | Baseline, 1 month, 3 months
  Change in creatinine levels
Safety Endpoint: Change in sodium levels | Baseline, 1 month, 3 months
  Change in sodium levels
Safety Endpoint: Change in potassium levels | Baseline, 1 month, 3 months
  Change in potassium levels

CONTACTS AND LOCATIONS:
Overall Officials: Emily Seto, PhD, Principal Investigator — University of Toronto
Locations (3):
- Canada (3):
  - North York General Hospital, North York, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware P, Dorai M, Ross HJ, Cafazzo JA, Laporte A, Boodoo C, Seto E. Patient Adherence to a Mobile Phone-Based Heart Failure Telemonitoring Program: A Longitudinal Mixed-Methods Study. JMIR Mhealth Uhealth. 2019 Feb 26;7(2):e13259. doi: 10.2196/13259. PMID 30806625
- [Background] Ware P, Ross HJ, Cafazzo JA, Laporte A, Gordon K, Seto E. Evaluating the Implementation of a Mobile Phone-Based Telemonitoring Program: Longitudinal Study Guided by the Consolidated Framework for Implementation Research. JMIR Mhealth Uhealth. 2018 Jul 31;6(7):e10768. doi: 10.2196/10768. PMID 30064970
- [Background] Ware P, Ross HJ, Cafazzo JA, Laporte A, Seto E. Implementation and Evaluation of a Smartphone-Based Telemonitoring Program for Patients With Heart Failure: Mixed-Methods Study Protocol. JMIR Res Protoc. 2018 May 3;7(5):e121. doi: 10.2196/resprot.9911. PMID 29724704
- [Background] Seto E, Leonard KJ, Cafazzo JA, Barnsley J, Masino C, Ross HJ. Mobile phone-based telemonitoring for heart failure management: a randomized controlled trial. J Med Internet Res. 2012 Feb 16;14(1):e31. doi: 10.2196/jmir.1909. PMID 22356799
- [Derived] Seto E, Ross H, Tibbles A, Wong S, Ware P, Etchells E, Kobulnik J, Chibber T, Poon S. A Mobile Phone-Based Telemonitoring Program for Heart Failure Patients After an Incidence of Acute Decompensation (Medly-AID): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jan 22;9(1):e15753. doi: 10.2196/15753. PMID 32012116